CLINICAL TRIAL: NCT04260230
Title: Remote Monitoring of Cancer Patients at Risk of Sepsis, a Pilot Study of Using Wearable Biosensors in Patients at High Risk of Chemotherapy Associated Neutropenic Sepsis
Brief Title: Remote Monitoring of Patients at Risk of Sepsis
Acronym: REACT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn without opening to recruitment
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: Isansys Lifecare LTD (Unknown); University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CFTSp172
Record Dates: First submitted 2020-01-14; First posted 2020-02-07 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Neutropenia, Febrile; Cancer; Sepsis
MeSH Terms: conditions — Febrile Neutropenia; Neoplasms; Sepsis

STUDY DESIGN:
Intervention Model Description: Single arm open label device tolerability study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lifetemp/Lifetouch sensors (Experimental): Participants will be asked to wear the sensors for six weeks. Data will be collected from the devices but will only be reviewed retrospectively and will not be used to alter participants care in any way.
  Interventions: Device: Lifetemp/Lifetouch sensors

INTERVENTIONS:
Device: Lifetemp/Lifetouch sensors — Wearing the devices for six weeks. Data only reviewed retrospectively.
  Other Names: Patient Status Engine

SUMMARY:
Chemotherapy is used to treat cancer in many thousands of patients per annum in the United Kingdom and millions worldwide.

Most chemotherapy suppresses bone marrow function and causes a low white cell count (neutropenia) which is a major cause of sepsis, a potentially fatal medical emergency. Best outcomes in sepsis result from early admission to hospital with the rapid start of antibiotics and supportive care. Currently, patients starting chemotherapy are told the importance of making contact with the hospital if they feel unwell or develop a high temperature. Despite this it is common for patients to delay telephoning the Cancer Centre "hot line" until after enduring many hours of symptoms and ultimately being admitted to hospital very unwell and sometimes in life threatening septic shock.

This proposal (REACT) seeks to invert the current model of care with the aim of improving patient outcomes whilst reducing costs. In this proof of concept pilot study the investigators aim to assess the feasibility of using remote wearable biosensors to record key physiological parameters (including respiratory rate, heart rate and temperature) and transmit this data centrally to The Christie. The investigators will also assess retrospectively whether perturbations in biosensor collected data correlate with clinical episodes of sepsis and if so develop bespoke clinical algorithms to identify patients displaying "red flags" for sepsis and guide response. Data collected by the sensors is at this stage only being reviewed retrospectively. Subsequent phases would involve recruiting larger number of patients to develop and test these algorithms with patients exhibiting 'red flags' for sepsis being contacted by the clinical team and taking appropriate action to facilitate assessment and treatment. The results of this study will determine whether working towards a randomised phase III trial comparing REACT with standard of care is an appropriate next step.

DETAILED DESCRIPTION:
This is a pilot, single arm, open label feasibility study. There will be no change in patient's clinical care. Physiological data will only be analysed retrospectively.

This is a single centre trial based in a large tertiary cancer centre that treats patients across all solid tumour and haematological malignancies. Patients will be recruited from lymphoma, haematology, lung and upper gastrointestinal disease groups.

All study procedures will be performed by a researcher who is appropriately trained and who has been delegated by the PI to undertake this activity (and this is clearly documented on the delegation log). No study specific procedures will take place prior to written informed consent being provided. Study Schedule (Main Study)

The main study will consist of the following visits:

Screening Visit 1 on day one of a cycle of planned standard of care chemotherapy. This visit will include application of the wearable biosensors and training in how to use the devices including cautions and safety advice. Participants will be provided with a diary to document any issues with the device or periods where the sensors are removed. This visit will include a standard of care review by the participant's direct care team. Visit 2 on day 1 of the next cycle of chemotherapy(3 weeks after Visit 1). This visit will include a review of any device related issues by the study team and completion of the relevant event checklist (version 1.0). The study diary will be reviewed. Used sensors will be collected and replacement sensors provided. The participant will be asked to complete an interim tolerability questionnaire. This visit will include a standard of care review by the participant's direct care team. Visit 3 on day 22 of either cycle 2, 3, or 4 (3 weeks after Visit 2). This visit will include a review of any device related issues by the study team and completion of the relevant event checklist (version 1.0). The study diary will be reviewed.

Used sensors will be collected. The participant will be asked to complete an end of study tolerability questionnaire.

This visit will include a standard of care review by the participant's direct care team.

Structured interview 1-4 weeks post Visit 3 with between 10 and 20 selected participants. This visit will take place either at the Christie in a private non-clinical space or via telephone, according to the participant's preference. The IRAS Form Reference: IRAS Version 5.13 Date: 9 DRAFT interview is expected to take approximately 30 minutes. This is a semi-structured interview which will follow the interview schema (version 1.0) Sub-study: This study will consist of one visit where the participant will be shown the sensors and explained how the investigators are intending to use them. They will then be asked to complete a questionnaire about how they feel about the sensors.

ELIGIBILITY:
Inclusion Criteria:

1. Participants are capable of giving informed consent
2. Male or female aged 18 or over
3. Diagnosis of malignancy including:

   * Lung cancer (including both small and non-small cell lung cancers)
   * Upper gastrointestinal malignancy
   * Haematological malignancy (lymphoma, leukaemia and myeloma)
4. Planned to commence chemotherapy OR undergoing chemotherapy in an outpatient setting as standard of care treatment with at least two cycles of treatment remaining.
5. Able to complete tolerability questionnaires.
6. Eastern Cooperative Oncology Group Performance Status <4
7. Life expectancy of greater than three months.

Exclusion Criteria:

1. Patients hospitalized at time of commencing chemotherapy
2. Pregnant patients
3. Patients unable to give informed consent
4. Presence of ulceration or pre-existing skin rash at site of device application (left precordium and axillae). If only one axilla affected this is not an exclusion criterion if patient is happy to apply temperature sensor to the other axilla.
5. Radiotherapy to the left chest wall either during or within the six months preceding the study. Plans for subsequent radiotherapy to commence after study completion are not an exclusion criterion. If only one axilla is within the planned radiotherapy field and patient is happy to apply temperature sensor to the other axilla this is not an exclusion criteria.
6. History of allergy or contact dermatitis to medical adhesives e.g sticking plasters, ECG electrodes.
7. Patients with pacemakers, implantable defibrillators or neurostimulators.
8. Patients who are currently receiving treatment as part of a clinical study or have had their end of treatment visit for another clinical study less than 30 days prior to Visit 1 are ineligible.
9. Patients who have planned foreign travel during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Device tolerability | Questionnaire at six weeks.
  Percentage of participants who answer 'agree' or 'strongly agree' on a five point Likert scale to the statement 'I would be happy to wear the sensors again if the data collected was being used to monitor my health during chemotherapy'. This statement is included in the questionnaires completed at the end of the device wearing period.

SECONDARY OUTCOMES:
Reliability of data transmission | Over six weeks of patients wearing devices.
  Reliable data transmission to central hospital system expressed as a percentage of total data points collected out of target data points collected.
Interim device tolerability | Questionnaire at three weeks.
  Percentage of participants who answer 'agree' or 'strongly agree' on a five point Likert scale to the statement 'I would be happy to wear the sensors again for the next three weeks'. This statement is included in the questionnaires completed after three weeks of wearing the device.
Semi-structured interviews | One to four weeks after completion of wearing the device.
  Device tolerability as assessed by semi-structured interviews.

OTHER OUTCOMES:
Correlation of physiological data with clinical events | Over 6 weeks of patients wearing devices.
  Exploratory analysis of sensor collected data with clinical episodes of infection. Sensor collected data includes heart rate, respiratory rate and temperature.

CONTACTS AND LOCATIONS:
Locations (1):
- The Christie NHS Foundation Trust, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No